CLINICAL TRIAL: NCT01414140
Title: Drug Use Investigation of Mirena
Brief Title: Mirena Post-marketing Surveillance in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15036; MIRENA (Other: Company Internal)
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Contraception
Keywords: Mirena, contraception
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Levonorgestrel IUS (Mirena, BAY86-5028)

INTERVENTIONS:
Drug: Levonorgestrel IUS (Mirena, BAY86-5028) — Women inserted Mirena for intrauterine contraception.

SUMMARY:
This study is a regulatory post-marketing surveillance in Japan, and it is a local prospective and observational study of women who are inserted Mirena for intrauterine contraception. The objective of this study is to assess safety and effectiveness of Mirena under real-life practice conditions. A total 550 patients will be recruited and followed for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Women who are inserted Mirena for intrauterine contraception Exclusion Criteria:
* Women who are contraindicated based on the product label

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population of this study is women who patients who are inserted Mirena for intrauterine contraception. The study is expected to collect data of 550 women.
Sampling Method: Non-Probability Sample
Enrollment: 567 (Actual)
Dates: Start 2007-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions and serious adverse events in women who are inserted Mirena | After Mirera insertion, up to 5 years
Incidence of adverse drug reactions, especially Pelvic inflammatory disease in women who are inserted Mirena | After Mirera insertion, up to 5 years

SECONDARY OUTCOMES:
Incidence of adverse drug reactions in subpopulation in a variety of baseline data (such as demographic data, concomitant disease) and duration of Mirena | After Mirera insertion, up to 5 years
Pregnancy rate | After Mirera insertion, up to 5 years
Released amount of Levonorgestrel [estimated from removed Mirena] | After Mirera insertion, up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Japan